CLINICAL TRIAL: NCT01149174
Title: Single Preoperative Intravesical Instillation of Electromotive Mitomycin-c for Primary Non-muscle Invasive Bladder Cancer: a Prospective Randomized Trial.
Brief Title: Preoperative Intravesical Electromotive Mitomycin-c for Primary Non-muscle Invasive Bladder Cancer
Acronym: EMDA/PRE-TUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Savino M. Di Stasi, Professor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EMDA/PRE-TUR/691836
Record Dates: First submitted 2009-11-18; First posted 2010-06-23 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Superficial Bladder Cancer
Keywords: intravesical chemotherapy; early single instillation; mitomycin-C; electromotive drug administration
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- transurethral resection alone (No Intervention): Patients with non-muscle invasive bladder cancer who underwent transurethral resection alone;
- intravesical mitomycin-C (Active Comparator): Patients with non-muscle invasive bladder cancer who underwent one intravesical instillation of mitomycin-C immediately after transurethral resection
  Interventions: Drug: Mitomycin-C 40 mg
- electromotive mitomycin-C (Experimental): Patients with non-muscle invasive bladder cancer who underwent single immediate intravesical instillation of electromotive mitomycin-C immediately before transurethral resection
  Interventions: Drug: Mitomycin-C 40 mg

INTERVENTIONS:
Drug: Mitomycin-C 40 mg — Intravesical instillation of Mitomycin-C
  Other Names: Mytomicin-C Kyowa Italiana Farmaceutici Milano
  Arms: electromotive mitomycin-C; intravesical mitomycin-C

SUMMARY:
Early single instillation of chemotherapy after TUR is recommended in the European Association of Urology Guidelines. Nevertheless, the procedure is suboptimal for patients with multiple tumors, sometimes is not tolerated and it can results in severe complications. In both laboratory and clinical studies, intravesical electromotive drug administration (EMDA) increases mitomycin-C (MMC) bladder uptake, resulting in an improved clinical efficacy in non-muscle invasive bladder cancer (NMIBC). The investigators will compare the effects of one immediate pre-TUR intravesical EMDA/MMC instillation with one immediate post-TUR intravesical passive diffusion MMC (PD/MMC) instillation and TUR alone in patients with NMIBC.

All eligible patients with primary NMIBC will be randomized into 3 groups who will undergo transurethral resection alone (TUR/alone); TUR plus single immediate postoperative instillation (immediately after TUR) of 40 mg PD/MMC with a dwell time of 60 minutes; or single immediate preoperative instillation (immediately before TUR) of 40 mg EMDA/MMC with 20 mA electric current for 30 minutes. Patients with intermediate and high risk NMIBC will undergo adjuvant intravesical therapy. The primary end points will be the recurrence rate and disease-free interval. All clinical analyses will be performed on an intent to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary histologically proven stage pTa-pT1 transitional-cell carcinoma of the bladder

Exclusion Criteria:

* Previous treatments with bacillus Calmette-Guerin, mitomycin-C, or with any other intravesical cytostatic agent
* Concomitant urothelial tumours of the upper urinary tract
* Previous or concomitant muscle-invasive (ie, stage T2 or higher) transitional-cell carcinoma of the bladder
* Bladder capacity less than 200 ml
* Untreated urinary-tract infection
* Disease of upper urinary tract
* Previous radiotherapy to the pelvis
* Other concurrent chemotherapy
* Treatment with radiotherapy-response or biological-response modifiers
* Other malignant diseases within 5 years of trial registration (except for basal-cell carcinoma)
* Pregnancy or nursing
* And psychological, familial or sociological factors that would preclude study participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 1994-01; Primary Completion 2003-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
disease-free interval and recurrence rate | recurrence assessed at 1 and 3 years from randomisation

SECONDARY OUTCOMES:
disease progression and overall and specific disease mortality | progression and mortality assessed at 5 years from randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Savino M Di Stasi, MD, PhD, Principal Investigator — "Tor Vergata" University, Rome, Italy
Locations (1):
- Dept. of Surgery, Tor Vergata University, Rome, Italy

REFERENCES:
- [Result] Di Stasi SM, Verri C, Capelli G, Brausi M , Leprini G, Casilio M, Zampa G. Single preoperative intravesical instillation of electromotive mitomycin-C for primary non- muscle-invasive bladder cancer: A prospective randomized trial. Journal of Clinical Oncology, 2010 ASCO Annual Meeting Proceedings. Vol 28, No 15 Suppl (May 20 Supplement), 2010: Abs # 4543.
- [Result] Di Stasi SM, Verri C, Capelli G, Brausi M, Leprini G, G Zampa, Stephen RL. Single preoperative intravesical instillation of electromotive mitomycin-C for primary non-muscle invasive bladder cancer: A randomized trial. The Journal of Urology, 2010 AUA Annual Meeting Proceedings. Vol 183, No. 4 Suppl (April Supplement), 2010: Abs #1346.
- [Result] Di Stasi SM, Valenti M, Verri C, Liberati E, Giurioli A, Leprini G, Masedu F, Ricci AR, Micali F, Vespasiani G. Electromotive instillation of mitomycin immediately before transurethral resection for patients with primary urothelial non-muscle invasive bladder cancer: a randomised controlled trial. Lancet Oncol. 2011 Sep;12(9):871-9. doi: 10.1016/S1470-2045(11)70190-5. Epub 2011 Aug 8. PMID 21831711